CLINICAL TRIAL: NCT03488823
Title: Evaluation of Effects of Flavonols on Endothelial Function and Hyperplasia of Intima After Endothelium Injury During Transradial Catheter.
Brief Title: Flavonols and Endothelial Injury
Acronym: Radialis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principle Investigator, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-012
Record Dates: First submitted 2018-02-15; First posted 2018-04-05 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Endothelial Dysfunction
Keywords: Endothelial Function; Flavonols; Intima Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young with Flavanol (Experimental): Young patients (< 45 years) will get twice daily from1 week vor catheterisation till one week after catheterisation drink with flavanols ( 2x400 mg Flavanols).
  Interventions: Dietary Supplement: with Flavanol
- Young without Flavanol (Placebo Comparator): Young patients (< 45 years) will get twice daily from1 week vor catheterisation till one week after catheterisation drink without flavanols .
  Interventions: Dietary Supplement: without Flavanol
- Old with Flavanol (Experimental): Old patients (>60 years) will get twice daily from1 week vor catheterisation till one week after catheterisation drink with flavanols ( 2x400 mg Flavanols).
  Interventions: Dietary Supplement: with Flavanol
- Old without Flavanol (Placebo Comparator): Young patients (>60 years) will get twice daily from1 week vor catheterisation till one week after catheterisation drink without flavanols.
  Interventions: Dietary Supplement: without Flavanol

INTERVENTIONS:
Dietary Supplement: with Flavanol — Patient will get twice daily drink rich on flavanols (400 mg) since one week before catheterization till one week after catheterization.
  Arms: Old with Flavanol; Young with Flavanol
Dietary Supplement: without Flavanol — Patient will get twice daily drink without flavanols since one week before catheterization till one week after catheterization.
  Arms: Old without Flavanol; Young without Flavanol

SUMMARY:
With increasing age, arterial endothelial cell function is impaired, which is associated with decreased regeneration response and increased intimal hyperplasia after endothelial injury. Dietary flavanols can reduce endothelial dysfunction acutely and chronically, but the exact mechanism is unknown. Recent studies suggest that flavanols may affect important endothelial regeneration response processes and possibly mediate long-term positive vascular effects. The aim of this study is to investigate age-dependent mechanisms of impaired endothelial regeneration and the influence of dietary flavanols on them. For this purpose, younger and old male patients, who are clinically indicated for elective transradial catheterization, will get periinterventional a test drink , which is rich on flavonols (800 mg flavanols daily), or control drink. Administration of drinks is randomized and double-blind. The test drinks should be given one week before the elective catheter examination until 1 week later. The endothelial regeneration is to be investigated as endothelium-dependent vasodilation non-invasively in the area of the puncture site on the forearm and by means of biomarkers in the blood. The endothelial function of the Arteria radialis will be measured with Flow Mediated Dilation (FMD) before and 24 h after catheterization. One month after catheterization patients undergo ultrasound examination of arteria radialis, to include structural vessel wall changes as intimal media thickness.

ELIGIBILITY:
Inclusion Criteria:

* planed catheterization, that has be done via Arteria radialis

Exclusion Criteria:

* acute infection (CRP>0.5 mg/dl)
* malignant diseases
* heart failure (NYHA III-IV)
* renal failure (GFR<60 ml/min)
* profoundly atrial fibrilation
* hypotension (≤100/60 mmHg)
* intolerance of nitroglycerin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Increase of Endothelial Function of Arteria radialis | week 2
  Change from Baseline Endothelial Function of Arteria radialis measured with Flow Mediated Dilation (FMD) after catheterization

SECONDARY OUTCOMES:
Degree of intimal Injury after Catheterization | 1 month
  Intimal Injury will be measured as intima media thickness with duplex sonography 1 month after catheterization

OTHER OUTCOMES:
Microvascular Function | 1 month
  Microvascular Function of Endothelium will be measured with Laser-Doppler Examination 1 month after catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Sansone, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Dusseldorf
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany